CLINICAL TRIAL: NCT03773107
Title: LCI-HEM-MYE-CRD-004 (MMRC-073 CARJAK): Phase I/II Study of Carfilzomib, Ruxolitinib, and Low Dose Dexamethasone for Carfilzomib-Refractory Multiple Myeloma
Brief Title: LCI-HEM-MYE-CRD-004 (MMRC-073 CARJAK): Study of CRD for Carfilzomib-Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Incyte Corporation (Industry); Multiple Myeloma Research Consortium (Network); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB00081612; 00031040 (Other: Advarra IRB); LCI-HEM-MYE-CRD-004 (Other: Atrium)
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Results first posted 2024-04-05 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
Keywords: Plasma Cell Neoplasms; Blood Malignancy
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — carfilzomib; ruxolitinib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I (Experimental): Cohort 1) 5mg ruxolitinib, Cohort 2) 10mg ruxolitinib, Cohort 3) 15mg ruxolitinib
  Interventions: Drug: Carfilzomib; Drug: Ruxolitinib; Drug: Dexamethasone
- Phase II (Other): Cohort A) non-responders to Phase I regimen, Cohort B) responders to Phase I regimen
  Interventions: Drug: Carfilzomib; Drug: Ruxolitinib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — Irreversible proteasome inhibitor
  Other Names: Kyprolis
Drug: Ruxolitinib — Oral JAK inhibitor
  Other Names: Jakafi
Drug: Dexamethasone — glucocorticoid

SUMMARY:
The primary objective of Phase I is to establish the maximum tolerated dose (MTD) of ruxolitinib in combination with carfilzomib and dexamethasone. The primary objective of phase II is to evaluate progression-free survival (PFS) at 4 months in multiple myeloma subjects who receive the combination treatment carfilzomib, dexamethasone, and ruxolitinib.

DETAILED DESCRIPTION:
This is an open-label, Phase I/II study of carfilzomib, ruxolitinib, and low-dose dexamethasone for carfilzomib-refractory multiple myeloma. Phase I is designed to evaluate overall maximum tolerated dose (MTD) of ruxolitinib in combination with carfilzomib and dexamethasone in the following cohorts: Cohort 1) 5mg ruxolitinib, Cohort 2) 10mg ruxolitinib, Cohort 3) 15mg ruxolitinib. Phase II is designed to evaluate 4-month progression-free survival (PFS) in the following cohorts: Cohort A) non-responders to Phase I regimen, Cohort B) responders to Phase I regimen. Up to 18 evaluable subjects will be enrolled in Phase I over approximately 12 months. An additional 30 evaluable subjects will be enrolled in Phase II over 24 months.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria:

1. Documented history of relapsed and/or refractory multiple myeloma with > 2 lines of therapy. One of the prior lines of therapy must have been a carfilzomib containing regimen with evidence of relapse or progression within the last 60 days of the carfilzomib containing regimen with a carfilzomib dose of at least 27 mg/m2. Carfilzomib containing regimen at the standard dose of 20/27 mg/m2 is acceptable.
2. Measurable disease, as defined by at least one of the following:

   1. Serum monoclonal protein level ≥0.5 g/dL for IgG, IgA, or IgM disease
   2. Urinary M-protein excretion of ≥200 mg over a 24-hour period
   3. Involved free light chain level ≥10 mg/dL, along with an abnormal free light chain ratio
3. Adequate bone marrow reserves, as defined by the following:

   1. Absolute neutrophil count (ANC) ≥1000 cells/mm3 within 1 week of the initiation of treatment
   2. Platelet count of ≥75 ,000 cells/mm3 for subjects who have bone marrow plasmacytosis of <50%, or ≥50,000 cells/mm3 for subjects who have bone marrow plasmacytosis of >50%
4. Adequate hepatic function, as defined by the following:

   1. Total bilirubin ≤ 2 times the upper limit of the institutional normal values
   2. Total AST and ALT ≤ 3 times the upper limit of the institutional normal values
5. Adequate renal function, as defined by the following: creatinine clearance (CrCl) ≥ 30 mL/min., as measured by a 24-hour urine collection, or estimated by the Cockcroft and Gault formula.
6. Adequate cardiac function defined as LVEF ≥ 40% by MUGA, echocardiogram or cardiac MRI.
7. Be 18-75 years of age
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
9. FOCBP and male subjects who are sexually active with FOCBP must agree to use two highly effective (as determined per the Investigator) methods of contraception during the study and for 30 days (female subjects) or for 90 days (male subjects) following the last dose of study treatment including a male condom.
10. Ability to understand and the willingness to sign a written informed consent document.
11. Recovered from all reversible acute toxic effects of prior therapy (other than alopecia) to ≤ Grade 1 or baseline.

Exclusion Criteria

Subjects must not meet any of the following criteria:

1. Non-secretory multiple myeloma
2. Known amyloidosis
3. Known POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
4. Clinically significant illness including, but not limited to the following: active systemic infection, uncontrolled hypertension (as defined by BP > 160/90), New York Heart Association Class III and IV heart failure, unstable angina pectoris, myocardial infarction within the past 6 months of consent, uncontrolled cardiac arrhythmia, or any other condition (including laboratory abnormalities) that, in the opinion of the Investigator, places the subject at unacceptable risk for adverse outcome if he/she were to participate in the study
5. Prior cerebrovascular accident with persistent neurologic deficit.
6. Psychiatric illness/social situations that would limit compliance with study treatment and requirements
7. Pregnant or breast feeding. Females of childbearing potential (FOCBP) must have a negative serum pregnancy test within the 7 days prior to study drug administration and a negative urine pregnancy test within the 3 days prior to the first study drug administration.
8. Known human immunodeficiency virus (HIV) infection
9. Active hepatitis B and/or hepatitis C infection
10. Currently active second malignancy, other than non-melanoma skin cancer and carcinoma in situ of the cervix, should not be enrolled. Subjects are not considered to have a currently active malignancy if they have completed therapy for a prior malignancy, are disease free from prior malignancies for >5 years, and are considered by their physician to be at less than 30% risk of relapse. In addition, subjects with basal cell carcinoma of the skin, superficial carcinoma of the bladder, carcinoma of the prostate with a current PSA value of <0.5 ng/mL, or cervical intraepithelial neoplasia will be eligible. Finally, subjects who are on hormonal therapy for a history of either prostate cancer or breast cancer may enroll, provided that there has been no evidence of disease progression during the previous three years.
11. Known history of allergy to Captisol® (a cyclodextrin derivative used to solubilize carfilzomib).
12. Contraindication to any of the required concomitant drugs or supportive treatments or intolerance to hydration due to preexisting pulmonary or cardiac impairment including pleural effusion requiring thoracentesis or ascites requiring paracentesis.
13. Known intolerance to carfilzomib.
14. Co-administration with strong CYP3A4 inhibitors (such as, but not limited to, boceprevir, clarithromycin, indinavir, itraconazole, ketoconazole, lopinavir/ritonavir, ritonavir, mibefradil, nefazodone, nelfinavir, posaconazole, saquinavir, telaprevir, telithromycin, voriconazole) as well as fluconazole (a dual inhibitor of CYP3A4 and CYP2C9).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2024-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shebli Atrash, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Karmanos Cancer Institute, Detroit, Michigan
  - Levine Cancer Institute, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The 10 participants who completed the Phase I component of the trial did not continue to the Phase II component of the trial. This is because the Phase II component of the trial did not open.
Groups:
- Phase I 5mg Ruxolitinib: Cohort 1) 5mg ruxolitinib
  Carfilzomib: Irreversible proteasome inhibitor
  Ruxolitinib: Oral JAK inhibitor
  Dexamethasone: glucocorticoid
- Phase I 10 mg Ruxolitinib: Cohort 2) 10mg ruxolitinib
  Carfilzomib: Irreversible proteasome inhibitor
  Ruxolitinib: Oral JAK inhibitor
  Dexamethasone: glucocorticoid
- Phase I 15 mg Ruxolitinib: Cohort 3) 15mg ruxolitinib
  Carfilzomib: Irreversible proteasome inhibitor
  Ruxolitinib: Oral JAK inhibitor
  Dexamethasone: glucocorticoid
Period: Overall Study
Arm/Group | Phase I 5mg Ruxolitinib | Phase II | Phase I 10 mg Ruxolitinib | Phase I 15 mg Ruxolitinib
Started | 5 | 0 (The Phase II component of this trial did not start.) | 4 | 3
Completed | 4 | 0 (The Phase II component of this trial did not start.) | 4 | 2
Not Completed | 1 | 0 | 0 | 1
Not completed — Participant currently on study and in follow up status. | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase I 10mg Ruxolitinib: Cohort 2) 10mg ruxolitinib
  Carfilzomib: Irreversible proteasome inhibitor
  Ruxolitinib: Oral JAK inhibitor
  Dexamethasone: glucocorticoid
- Phase I 15 mg Ruxolitibin: Cohort 3) 15mg ruxolitinib
  Carfilzomib: Irreversible proteasome inhibitor
  Ruxolitinib: Oral JAK inhibitor
  Dexamethasone: glucocorticoid
- Total: Total of all reporting groups
Arm/Group | Phase II | Phase I 5mg Ruxolitinib | Phase I 10mg Ruxolitinib | Phase I 15 mg Ruxolitibin | Total
Number analyzed (Participants) | 0 | 5 | 4 | 3 | 12
Age, Categorical [Count of Participants; unit: Participants] — Population: Note: the sum of the number of participants who started in the Age subgroups add up to the total number of participants who started for each of the respective ruxolitinib dose levels.
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 0 | 2 | 2 | 1 | 5
    >=65 years | 0 | 3 | 2 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Note: the sum of the number of participants who started in the Sex subgroups add up to the total number of participants who started for each of the respective ruxolitinib dose levels.
  Participants
    Female | 0 | 0 | 2 | 1 | 3
    Male | 0 | 5 | 2 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Note: the sum of the number of participants who started in the Ethnicity subgroups add up to the total number of participants who started for each of the respective ruxolitinib dose levels.
  Participants
    Hispanic or Latino | 0 | 1 | 0 | 0 | 1
    Not Hispanic or Latino | 0 | 4 | 4 | 3 | 11
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 2
  White | 0 | 3 | 3 | 3 | 9
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants] — Population: Note: the sum of the number of participants who started in the Region subgroups add up to the total number of participants who started for each of the respective ruxolitinib dose levels.
  participants
    United States |  | 5 | 4 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT)
Description: DLTs will be determined for each subject as a binary variable indicating whether or not the subject experienced a DLT during Cycle 1
Time Frame: 28 days
Population: Participants who are DLT evaluable
Measure: Number; unit: participants
Groups:
- Phase I 5 mg Ruxolitinib: Cohort 1) 5mg ruxolitinib
  Carfilzomib: Irreversible proteasome inhibitor
  Ruxolitinib: Oral JAK inhibitor
  Dexamethasone: glucocorticoid
Arm/Group | Phase I 5 mg Ruxolitinib | Phase I 10 mg Ruxolitinib | Phase I 15 mg Ruxolitinib
Number analyzed (Participants) | 3 | 3 | 2
participants | 0 | 0 | 1

2. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response will be determined for each subject as a binary variable indicating whether or not the subject achieved a best overall response of PR or better as per the IMWG criteria
Time Frame: Approximately 180 days after treatment start (disease assessment occurred after every 28-day cycle)
Population: Participants who initiate protocol-directed therapy and have measurable disease at baseline.
Measure: Number; unit: participants
Arm/Group | Phase I 5mg Ruxolitinib | Phase I 10 mg Ruxolitinib | Phase I 15 mg Ruxolitibin
Number analyzed (Participants) | 5 | 4 | 3
participants | 0 | 2 | 1

3. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit will be determined for each subject as a binary variable indicating whether or not the subject achieved a best overall response of minimal response (MR) or better as determined by the IMWG criteria
Time Frame: Approximately 180 days after treatment start (disease assessment occurred after every 28-day cycle)
Population: Participants who initiate protocol-directed therapy and have measurable disease at baseline.
Measure: Number; unit: participants
Groups:
- Phase I 5m Ruxolitinib: Cohort 1) 5mg ruxolitinib
  Carfilzomib: Irreversible proteasome inhibitor
  Ruxolitinib: Oral JAK inhibitor
  Dexamethasone: glucocorticoid
Arm/Group | Phase I 5m Ruxolitinib | Phase I 10 mg Ruxolitinib | Phase I 15 mg Ruxolitinib
Number analyzed (Participants) | 5 | 4 | 3
participants | 1 | 2 | 1

4. Secondary Outcome: Disease Control Rate
Description: Disease control will be determined for each subject as a binary variable indicating whether or not the subject achieved a disease response or stable disease for greater than or equal to 8 weeks
Time Frame: Approximately 180 days after treatment start (disease assessment occurred after every 28-day cycle)
Population: Number of participants who achieved a disease response of stables disease or better and maintained the response for at least 8 weeks.
Measure: Number; unit: participants
Arm/Group | Phase I 5mg Ruxolitinib | Phase I 10 mg Ruxolitinib | Phase I 15 mg Ruxolitinib
Number analyzed (Participants) | 5 | 4 | 3
participants | 3 | 3 | 1

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the duration of time from the initiation of study treatment with ruxolitinib to first occurrence of either progressive disease or death without progressive disease.
Time Frame: approx. 5 years
Population: All participants who initiate study treatment.
Measure: Median (Inter-Quartile Range); unit: months
Groups:
- Phase I 15mg Ruxolitinib: Cohort 3) 15mg ruxolitinib
  Carfilzomib: Irreversible proteasome inhibitor
  Ruxolitinib: Oral JAK inhibitor
  Dexamethasone: glucocorticoid
Arm/Group | Phase I 5mg Ruxolitinib | Phase I 10mg Ruxolitinib | Phase I 15mg Ruxolitinib
Number analyzed (Participants) | 5 | 4 | 3
months | 3.0 [1.8 to 3.2] | 6.1 [2.6 to 8.3] | 10.6 [1.3 to 10.6]

6. Secondary Outcome: Time to Best Response
Description: Time to best response will be defined as the time from initiation of ruxolitinib treatment to the time of best objective status assessment of response.
Time Frame: Approximately 180 days after treatment start (disease assessment occurred after every 28-day cycle)
Population: Time to best response calculated only for participants who achieved a PR or better.
Measure: Median (Full Range); unit: months
Arm/Group | Phase I 5 mg Ruxolitinib | Phase I 10 mg Ruxolitinib | Phase I 15 mg Ruxolitinib
Number analyzed (Participants) | 0 | 2 | 1
months |  | 3.2 [1.8 to 4.6] | 2.1 [2.1 to 2.1]

7. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the duration from initiation of ruxolitinib treatment to the date of death from any cause.
Time Frame: approx. 5 years
Population: All participants who initiate study treatment.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Phase I 5mg Ruxolitinib | Phase I 10mg Ruxolitinib | Phase I 15mg Ruxolitinib
Number analyzed (Participants) | 5 | 4 | 3
months | 16.1 [15.9 to 23.5] | 11.2 [5.9 to 13.1] | 10.6 [1.3 to 19.4]

8. Secondary Outcome: Time to Progression
Description: Time to progression (TTP) is defined as the duration of time from the initiation of study treatment with ruxolitinib to first occurrence of either progressive disease or death.
Time Frame: approx. 5 years
Population: All participants who initiate study treatment.
Measure: Mean (Inter-Quartile Range); unit: months
Arm/Group | Phase I 5mg Ruxolitinib | Phase I 10mg Ruxolitinib | Phase I 15mg Ruxolitinib
Number analyzed (Participants) | 5 | 4 | 3
months | 3.0 [1.8 to 3.2] | 8.3 [4.0 to 8.3] | 10.6 [10.6 to 10.6]

9. Secondary Outcome: Duration of Response
Description: Duration of response will be defined as the time from first objective status assessment of response to the time of first documented disease progression or death.
Time Frame: approx. 5 years
Population: Duration of best response calculated only for participants who achieved a PR or better.
Measure: Median (Full Range); unit: months
Arm/Group | Phase I 5mg Ruxolitinib | Phase I 10 mg Ruxolitinib | Phase I 15mg Ruxolitinib
Number analyzed (Participants) | 0 | 2 | 1
months |  | 4.8 [2.2 to 7.4] | 8.5 [8.5 to 8.5]

ADVERSE EVENTS:
Time Frame: Approximately 5 years
Arm/Group | Phase I 5 mg Ruxolitinib | Phase I 10 mg Ruxolitinib | Phase I 15 mg Ruxolitinib
All-Cause Mortality (participants affected / at risk) | 4/5 | 3/4 | 2/3
Serious Adverse Events (participants affected / at risk) | 4/5 | 3/4 | 1/3
Other Adverse Events (participants affected / at risk) | 5/5 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I 5 mg Ruxolitinib (N=5) | Phase I 10 mg Ruxolitinib (N=4) | Phase I 15 mg Ruxolitinib (N=3)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Septic shock.
Acute kidney injury (Renal and urinary disorders) | 0 | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
ALT increase (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Pneumonia.
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) — Death.
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I 5 mg Ruxolitinib (N=5) | Phase I 10 mg Ruxolitinib (N=4) | Phase I 15 mg Ruxolitinib (N=3)
Anemia (Blood and lymphatic system disorders) | 4 (9) | 4 (26) | 2 (10)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
ALT increase (Investigations) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
AST increase (Investigations) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — It is unknown whether the chest pain was of cardiac origin or not.
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 3 (3) | 1 (3) | 1 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 0 (0) — Intermittent dyspnea (1 event). Dyspnea on exertion (1 event).
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) — Ear stuffiness.
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0) — Bilateral lower extremities.
Ejection fraction decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Enterocolitis (c diff).
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (2) | 0 (0) — Eyelid stye.
Fatigue (General disorders) | 2 (2) | 2 (2) | 0 (0) — Due to disease progression (1 event).
Fever (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Right sided weakness.
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) — Headaches (intermittent), 1 event.
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (4) — Pneumonia (2 events).
Malaise (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Muscle cramps and twitching.
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) — Tingling in skin while showering (1 event), left sided gaze (1 event).
Neutrophil count decreased (Investigations) | 2 (3) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) — Achy all over body (1 event).
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (20) | 3 (9) | 2 (7)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — Altered mental state.
Purpura (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Shortness of breath.
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Squamous Cell Carcinoma (left temple).
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Abscess buttocks.
Soar throat (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) — Urinary frequency/retention (1 event), urinating at night, specifically (1 event).
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Weight loss (Investigations) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The Phase II part of the trial did not open to enrollment. The MTD was not identified in the Phase I part of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT03773107/Prot_SAP_001.pdf
  • Informed Consent Form (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT03773107/ICF_000.pdf